CLINICAL TRIAL: NCT04130737
Title: The PQ Bypass Pivotal IDE Intra-arterial Stent Graft Study for Occlusive and Re-stenotic Fem-pop Revascularization - 2 Trial: TORUS 2
Brief Title: TORUS 2 IDE Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Collaborators: Syntactx (Network); PQ Bypass, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 227
Record Dates: First submitted 2019-10-10; First posted 2019-10-17 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Artery Disease; Superficial Femoral Artery; Popliteal Artery; Stent Graft
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TORUS Stent Graft System (Experimental): The TORUS Stent Graft System (SGS) is comprised of a Stent Graft (SG) and a Stent Graft Delivery System (SGDS).
  Interventions: Device: TORUS Stent Graft System

INTERVENTIONS:
Device: TORUS Stent Graft System — The TORUS Stent Graft is an intravascular prosthesis intended to improve blood flow in the area in which it is implanted and the TORUS Stent Graft Delivery System is a standard pin-and-pull delivery system used to implant the SG in the desired area. Use of the TORUS Stent Graft allows for improving blood flow in the peripheral vasculature.
  Other Names: TORUS Stent Graft; PQ Bypass™ Stent Graft System

SUMMARY:
The primary objective of the TORUS 2 IDE Clinical Study is to evaluate the safety and effectiveness of the TORUS Stent Graft System in the treatment of obstructive atherosclerotic lesions of the native SFA or the superficial femoral and/or proximal popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female, with age > 18 and ≤ 90 years at date of enrollment.
2. Patient provides written informed consent before any study-specific investigations or procedures.
3. Patient is willing to undergo all follow-up assessments according to the specified schedule over 36 months.
4. Patient is a suitable candidate for angiography and endovascular intervention and, if required, is eligible for standard surgical repair.
5. Patient has symptomatic peripheral arterial disease (PAD) of the lower extremities requiring intervention to relieve de novo obstruction or occlusion or restenosis of the native femoropopliteal artery.
6. Patient has PAD classified as Rutherford classification 2, 3 or 4.
7. Patient has documented PAD by either (i) a resting ankle-brachial index (ABI) of ≤ 0.90 (or ≤ 0.75 after exercise of the target limb). Resting toe brachial index (TBI) is performed only if unable to reliably assess ABI. TBI must be <0.70; or (ii) Normal ABI with angiographic, ultrasound, MRA, or CT evidence of ≥ 60% diameter stenosis.
8. Patient has single or multiple stenotic, restenotic or occlusive lesions within the native femoropopliteal artery ("target lesions") that can be crossed with a guidewire and fully dilated.
9. Single target lesion must be covered by a single stent. Tandem target lesions are considered a single continuous lesion if the gap between lesions is ≤ 5 cm and > 30% diameter stenosis between the lesion(s).
10. Target lesion(s) eligible for treatment under the protocol are at least least 3 cm above the bottom of the femur.
11. Target lesion(s) reference vessel diameter is between 5.0 mm and 6.7 mm by operator's visual estimate.
12. Target lesion measures ≥ 80 mm to ≤ 180 mm in overall length, with ≥ 60% diameter stenosis by operator's visual estimate. Tandem target lesions are considered a single continuous lesion if the gap between lesions is ≤ 5 cm and > 30% diameter stenosis between the lesion(s).
13. Patient has a patent popliteal artery (no stenosis ≥ 50%) distal to the treated segment.
14. Patient has at least one patent infrapopliteal vessel (< 50% stenosis) with run-off to the ankle.

Exclusion Criteria:

1. Patient is unable or is unwilling to comply with the procedural requirements of the study protocol or will have difficulty in complying with the requirements for attending follow-up visits.
2. Patient has a comorbidity that in the investigator's opinion would limit life expectancy to less than 24 months.
3. Patient has any planned major surgical procedure (including any amputation of the target limb) within 30 days after the index procedure for this study.
4. Patient has a target vessel that has been treated with any type of surgical procedure prior to enrollment.
5. Patient has a target vessel that has been treated with bypass surgery.
6. Patient has PAD classified as Rutherford classification 0, 1, 5 or 6.
7. Patient has known or suspected active systemic infection at the time of enrollment.
8. Patient has a known coagulopathy or has bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter or INR (international normalized ratio) >1.8.
9. Patient has a stroke diagnosis within three months prior to enrollment.
10. Patient has a history of unstable angina or myocardial infarction within 60 days prior to enrollment.
11. Patient has a contraindication to antiplatelet, anticoagulant or thrombolytic therapies.
12. Patient has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-medicated.
13. Patient has known allergy to titanium, nickel or tantalum (does not include mild contact dermatitis due to nickel allergy).
14. Patient has received thrombolysis within 72 hours prior to the index procedure.
15. Patient has acute or chronic renal disease (e.g., as measured by a serum creatinine of > 2.5 mg/dL or > 220 μmol/L or GFR < 30 ml/min), or on peritoneal or hemodialysis.
16. Patient requiring coronary intervention within seven days prior to enrollment.
17. Patient is pregnant or breast-feeding.
18. Patient is participating in another research study involving an investigational product (pharmaceutical, biologic or medical device).
19. Patient has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
20. Patient has significant disease or obstruction (≥ 50%) of the inflow tract that has not been successfully treated at the time of the index procedure (success measured as ≤ 30% residual stenosis, without complication).
21. Patient has no patent (≥ 50% stenosis) outflow vessel providing run-off to the ankle.
22. There is a lack of full expansion in the predilatation balloon.
23. Evidence of aneurysm or acute thrombus in target vessel.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Freedom from a Major Adverse Event (MAE) | 30 days
  An MAE is defined as all-cause death, target limb major amputation and clinically-driven target lesion revascularization (CD-TLR)
Primary Patency | 12 months
  Primary patency is defined as the absence of clinically-driven target lesion revascularization (CD-TLR) and absence of recurrent target lesion diameter stenosis >50% by duplex ultrasound with a peak systolic velocity ratio of >2.5.

SECONDARY OUTCOMES:
Technical Success | At the time of the index procedure
  Technical success is defined as the ability to cross and dilate the lesion to achieve residual stenosis of ≤30%
Procedural Success | Within 24 hours of the procedure
  Procedural Success is defined as technical success with out any MAEs.
Major Adverse Event (MAE) Rate | 12 months
  Composite rate of all-cause death, target limb major amputation and clinically-driven target lesion revascularization (CD-TLR).
Patency Rate | Through 36 months
  Absence of CD-TLR and absence of recurrent target lesion diameter stenosis >50% by duplex ultrasound with a peak systolic velocity ratio of >2.5.
Assisted Primary Patency Rate | Through 36 months
  Revascularization of non-occlusive (<99%) stenosis within the stent graft or immediately above or below the treated arterial segment (end of the graft and 1cm of artery beyond) with less than 50% residual stenosis.
Secondary Patency Rate | Through 36 months
  Revascularization of occlusion (100%) within the stent graft or immediately above or below the treated arterial segment (end of the graft and 1cm of artery beyond) with less than 50% residual stenosis.)
Alternative Patency Rate | Through 36 months
  Patency of target vessel based on systolic velocity ratio ≤ 2.0 and absence of CD-TLR.
Walking Improvement Questionnaire (WIQ) Assessment | From procedure to 1, 6 and 12 months
  Assessment of walking improvement
Quality of Life Assessment by the EQ5D | From procedure to 1, 6 and 12 months
  Assessment of improved quality of life
Clinically Driven Target Lesion Revascularization | Through 36 months
Target Vessel Revascularization | Through 36 months
Major Amputation on Target Limb | Through 36 months
Stent Fracture Rate | 12 months
  Stent fracture rate using VIVA definitions
Change in Ankle-Brachial Index | From procedure through 36 months
Change in Toe Pressures | From procedure through 36 months
Change in Rutherford Clinical Classification | From procedure through 36 months
Adverse Event Rate | Through 36 months

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Southwest CVA, Mesa, Arizona
  - Vascular Heart & Lung Associates, Mesa, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Yuma Cardiology Associates, Yuma, Arizona
  - Arkansas Heart, Little Rock, Arkansas
  - Bay Area Vein & Vascular Institute, Burlingame, California
  - UCSF, San Francisco, California
  - Rocky Mountain Regional VAMC, Aurora, Colorado
  - The Vascular Experts, Darien, Connecticut
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Palm Vascular Centers, Miami Beach, Florida
  - Coastal Vascular & Interventional, Pensacola, Florida
  - Florida Cardiology, Winter Park, Florida
  - AMITA Health, Elk Grove, Illinois
  - MedStar Health Research Insitute, Hyattsville, Maryland
  - McLaren Bay Region, Bay City, Michigan
  - Michigan Vascular Center, Flint, Michigan
  - Eastlake Cardiovascular, Roseville, Michigan
  - Northern Mississippi Medical Center, Tupelo, Mississippi
  - Columbia University Medical Center, New York, New York
  - Novant Health, Charlotte, North Carolina
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - The Lindner Center for Research & Education, Cincinnati, Ohio
  - Naadi, Oklahoma City, Oklahoma
  - The Miriam Hospital, Providence, Rhode Island
  - Prisma Health, Greenville, South Carolina
  - North Central Heart, Sioux Falls, South Dakota
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Texas Tech, Lubbock, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Bellin Hospital, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No